CLINICAL TRIAL: NCT00189852
Title: Supporting Care and Independence at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barnsley Hospital (Other)
Collaborators: Engineering and Physical Sciences Research Council, UK (Other); Imperial College London (Other); University College, London (Other); University of Dundee (Other); Anchor Trust (Other); Thomas Pocklington Trust (Other); Tunstall (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EPSRC Grant No. GR/S29058/01
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: Telecare; chronic; older people; heart failure
MeSH Terms: conditions — Heart Failure; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docobo (Experimental): telemonitoring at home system for heart failure
  Interventions: Device: Chronic heart failure monitoring system; Device: Lifestyle monitoring system
- Control (No Intervention): No telemonitoring system in place

INTERVENTIONS:
Device: Chronic heart failure monitoring system
  Arms: Docobo
Device: Lifestyle monitoring system
  Arms: Docobo

SUMMARY:
The primary objective of this project is to investigate whether, in a pilot randomised controlled trial, the use of telecare (remote monitoring) technologies reduces the frequency of hospital admissions for people with chronic heart failure (CHF) and to inform the design of a larger randomised controlled trial of telecare for CHF.

Secondary objectives are:

1. To investigate whether there are benefits to users
2. To understand the impact on carers in terms of carer stress
3. To investigate whether there are benefits to the NHS and other statutory provisions
4. To investigate which users receive the greatest benefits
5. To inform whether remote monitoring of CHF patients should be provided as part of hospital discharge for a set period of time or whether it should be provided long term and be used in a preventative manner
6. To investigate whether CHF episodes can be detected and predicted based on lifestyle changes
7. To determine whether lifestyle monitoring equipment can be correlated with the information from the CHF monitoring system to determine the potential to detect deteriorating health.

DETAILED DESCRIPTION:
The 2004 Department of Health publication "Improving Chronic Disease Management" highlights that: 17.5 m adults in the UK may be living with a chronic disease; Around 80% of GP admissions relate to chronic disease; Patients with a chronic disease or complications use over 60% of hospital beds. Evidence from the US suggests that people with chronic conditions consume 78% of all health spending. The NHS modernisation agency has suggested that patients with chronic diseases should, in the future, no longer end up in acute beds when they could be treated in a community setting, or supported at home.

Chronic heart failure (CHF) is a major chronic disease which has been recognised in the UK with a National Service Framework (NSF) for Coronary Heart Disease. In industrialised countries it affects 1% of the population on average and 10% at 70 years of age. It accounts for 5 per cent of all medical admissions to the hospital (120,000 hospital admissions annually) costing an estimated £360 million to the NHS with 6,000 deaths each year from CHF.

The disease has a poor prognosis as within 5 years of diagnosis there is a 50% mortality, and many debilitating, costly and unplanned hospital admissions. Indeed, as many as 50% of patients are readmitted within 3 months of initial discharge. It has been suggested that up to 50% of hospital admissions for heart failure are preventable.

Telecare proposes an earlier diagnosis and with more appropriate and timely use of drugs this can increase patient survival and their quality of life. A weight gain of just a few pounds can signal that a chronic heart failure patient is retaining fluid, for example. If caught early enough, the patient may be able to take medication or otherwise manage the problem at home, rather than having to be hospitalised which improves care and saves money. There is extensive evidence that hospitalisation rates in patients with heart failure can be substantially reduced by improved patient education, patient self monitoring of weight, and rapid response to early signs of clinical deterioration. Telehealth interventions for CHF have tended to be based on devices asking specific questions with answers being entered by users. The information provided is then often supplemented with data from weighing scales and blood pressure monitors, with this being forwarded through the telephone system to a central sever. Here medical staff review the data and respond to patients with increasing risk. Automated software is also becoming available that can highlight to practitioners when a certain patient is outside of practitioner defined parameters or is not using their equipment regularly.

Lifestyle monitoring systems, using movement detectors and magnetic proximity switches on fridge and entry doors, can generate a profile of the user's lifestyle. Deviations from the normal profile can result in an alert being generated.

Correlations between both health and lifestyle strategies have not been conducted and this trial provides this opportunity.

Within the realms of this research study the lifestyle monitoring system will not be utilising the 'alert' system. It will purely be in a data gathering mode.

ELIGIBILITY:
Inclusion Criteria:

* Participants identified as having chronic heart failure
* Over the age of 60
* New York Heart Association (NYHA) functional classification 2, 3, or 4.

Exclusion Criteria:

* Ejection fraction more than 40%
* Under the age of 60
* Class 1 as determined by the NYHA

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Different number of hospital admissions between groups

SECONDARY OUTCOMES:
Benefits to users
Impact on carers

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hawley, Principal Investigator — Barnsley Hospital NHS Foundation Trust
Locations (1):
- Barnsley Hospital NHS Foundation Trust, Barnsley, Yorkshire, United Kingdom